CLINICAL TRIAL: NCT03025828
Title: Changes in Autoreactive Memory B Cells as Biomarker of Response to Adrenocorticotropic Hormone in Patients With Membranous Nephropathy
Brief Title: Adrenocorticotropic Hormone in Membranous Nephropathy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Principal Investigator, Paolo Cravedi, Assistant Professor, Nephrology, Icahn School of Medicine at Mount Sinai
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GCO 16-2402
Record Dates: First submitted 2017-01-17; First posted 2017-01-20 (Estimated); Results first posted 2022-08-15 (Actual); Last update posted 2022-08-15 (Actual); Status verified 2022-07

CONDITIONS: Membranous Nephropathy
Keywords: Membranous nephropathy; adrenocorticotropic hormone; ACTH; proteinuria; glomerulonephritis
MeSH Terms: conditions — Glomerulonephritis, Membranous; Proteinuria; Glomerulonephritis | interventions — Adrenocorticotropic Hormone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Acthar (Experimental): Acthar will be administered subcutaneously (SC) 80 units for the first week and then 80 units twice weekly
  Interventions: Drug: ACTHar

INTERVENTIONS:
Drug: ACTHar — for 6 months
  Other Names: ACTH; Acthar Injectable Product; Repository corticotropin injection; RCI; Acthar® Gel

SUMMARY:
The purpose of this study is to evaluate the effect of adrenocorticotropic hormone (ACTH, Acthar) on the loss of proteins in the urine (proteinuria) in patients with membranous nephropathy. Acthar is a hormone that stimulates steroid production from small glands above the kidneys. It has direct protective effects on the kidney and is currently approved by the FDA to treat kidney disorders associated with proteins in the urine, but the mechanisms of action are not entirely understood and will be studied in the present trial.

DETAILED DESCRIPTION:
Patients with membranous nephropathy and nephrotic syndrome will be treated with ACTH for 6 months. Proteinuria remission at 12 months will be the primary endpoint. Different biomarkers including anti-PLA2R autoantibodies, circulating regulatory T cells, and autoreactive memory B cells will be serially measured to identify predictors of response to therapy.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 70 years
* Free of immunosuppression for at least 3 months
* Capability of understanding the purpose of the study
* Written informed consent

Exclusion Criteria:

* Epidermal growth factor receptor (eGFR) < 30ml/min/1.73m2
* Kidney Transplant
* Secondary MN (defined on the basis of clinical criteria)
* Type 1 or Type 2 diabetes mellitus (prior diagnosis of gestational diabetes mellitus is not an exclusion)
* History of previous use of Acthar for treatment of nephrotic syndrome
* Prior sensitivity to Acthar or other porcine protein products
* Contraindication to Acthar per Prescribing Information
* Planned treatment with live or live attenuated vaccines once enrolled in the study
* More than three previous treatment regiments
* Participation to other clinical trials over the previous 12 months
* History of cancer, except carcinoma in situ and treated basal and squamous cell carcinomas
* Pregnancy
* Lactation
* Current substance abuse
* Any clinically relevant condition that might affect study participation and/or study results

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2018-03-19 (Actual); Primary Completion 2020-12-16 (Actual); Study Completion 2020-12-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paolo Cravedi, MD, PhD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Enrollment from March 2018 and June 2019
Groups:
- Acthar: Acthar will be administered subcutaneously (SC) 80 units for the first week and then 80 units twice weekly for 6 months
Period: Overall Study
Arm/Group | Acthar
Started | 5
Completed | 4
Not Completed | 1
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Groups:
- Acthar: Acthar administered subcutaneously (SC) 80 units for the first week and then 80 units twice weekly for 6 months of treatment with a cumulative dose exposure of 3,920 units.
Arm/Group | Acthar
Number analyzed (Participants) | 4
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.75 (8.098)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 4
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Serum albumin [Mean (Standard Deviation); unit: g/dL] | 3 (1.01)
Serum creatine [Mean (Standard Deviation); unit: mg/dL] | 0.965 (0.118)
Negative for Anti-PLA2R Ab [Count of Participants; unit: Participants] — Threshold for anti-PLA2R Ab positivity is 19.9 RU/mL.
  Participants | 4
Urine protein/creatinine ratio (P/C) [Mean (Standard Deviation); unit: g/g] | 6.173 (3.545)
Number of Participants with previous treatment [Count of Participants; unit: Participants] — Participants who had previously received treatment with steroids, alkylating agents, calcineurin inhibitors, and/or rituximab.
  Participants | 2

OUTCOME MEASURES:

1. Primary Outcome: Change in Proteinuria
Description: Change in proteinuria at baseline versus after 12 months of treatment as measured by urine protein/creatinine ratio
Time Frame: baseline and 12 months
Measure: Median (Inter-Quartile Range); unit: ratio
Arm/Group | Acthar
Number analyzed (Participants) | 4
ratio
  baseline | 4.56 [4.41 to 6.32]
  12 months | 1.36 [1.1 to 1.78]

2. Secondary Outcome: Number of Participants With Complete or Partial Remission
Description: Complete (proteinuria reduction <500mg/24h) or partial (urinary protein excretion (P/C) <3.0 g/g (with at least 50% reduction versus baseline) in at least two consecutive visits) remission.
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Acthar
Number analyzed (Participants) | 4
Participants
  complete remission | 0
  partial remission | 4

3. Secondary Outcome: Change in Serum Albumin
Description: Change in serum albumin from baseline
Time Frame: baseline 6 months, 12 months
Measure: Median (Inter-Quartile Range); unit: g/dl
Arm/Group | Acthar
Number analyzed (Participants) | 4
g/dl
  baseline and 6 months | 3.0 [2.03 to 3.98]
  baseline and 12 months | 3.65 [3.4 to 4.2]

4. Secondary Outcome: Estimated Glomerular Filtration Rate (GFR)
Description: GFR measures kidney function.
Time Frame: baseline and 12 months
Measure: Median (Inter-Quartile Range); unit: mL/min
Arm/Group | Acthar
Number analyzed (Participants) | 4
mL/min
  baseline | 90.5 [74.74 to 103.3]
  12 months | 80.5 [66.0 to 101.8]

5. Secondary Outcome: Number of Anti-PLA2R Memory B Cells
Description: Number of anti-PLA2R memory B cells
Time Frame: 12 months
Population: Data not collected
Arm/Group | Acthar
Number analyzed (Participants) | 0

6. Secondary Outcome: Anti-PLA2R Antibodies Levels
Description: blood levels
  Number of anti-PLA2R memory B cells
Time Frame: 12 months
Population: Data not collected
Arm/Group | Acthar
Number analyzed (Participants) | 0

7. Secondary Outcome: Change in CD4+CD25+CD127low T Regulatory Cells/CD4+ T Cell Ratio
Description: blood levels - one single cell subset identified by different markers
Time Frame: baseline and 12 months
Measure: Median (Inter-Quartile Range); unit: ratio
Arm/Group | Acthar
Number analyzed (Participants) | 4
ratio
  Baseline | 0.04 [0.03 to 0.06]
  12 Months | 0.12 [0.08 to 0.14]

ADVERSE EVENTS:
Time Frame: 12 months
Arm/Group | Acthar
All-Cause Mortality (participants affected / at risk) | 0/4
Serious Adverse Events (participants affected / at risk) | 0/4
Other Adverse Events (participants affected / at risk) | 0/4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-07-16): https://cdn.clinicaltrials.gov/large-docs/28/NCT03025828/Prot_SAP_000.pdf